CLINICAL TRIAL: NCT02415192
Title: A Multicenter, Prospective Observational Study to Evaluate the Safety and Efficacy for Levacalm Tab. Versus Valsartan/Amlodipine Combination Therapy in Patient With Essential Hypertension
Brief Title: Observational Study to Evaluate the Safety and Efficacy for Levacalm Tab. Versus Valsartan/Amlodipine Combination Therapy in Essential Hypertension Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-ZVOS001
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Lower Leg Edema; Orthostatic Hypertension
Keywords: safety data; hypertension therapy
MeSH Terms: interventions — Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients treated with Levacalm: In this group, the patients will be enrolled treated with Levacalm tab. as an anti-hypertensive drug.
  The number of this group will be double than the control group to get more information about safety and efficacy.
  Interventions: Drug: Levacalm
- Patients treated with Valsartan/amlodipine: In this group, the patients will be enrolled treated with Valsartan/amlodipine combination drug as an anti-hypertensive drug.
  Interventions: Drug: Valsartan/amlodipine

INTERVENTIONS:
Drug: Levacalm
  Groups: Patients treated with Levacalm
Drug: Valsartan/amlodipine
  Groups: Patients treated with Valsartan/amlodipine

SUMMARY:
Levacalm Tab. was approved in Jul 2013 by MFDS in South Korea. Levacalm Tab. is combination drug of Valsartan as an angiotensin II receptor blocker and Lercanidipine as a Calcium channel blocker. It is a new drug of combination of Valsartan and Lercanidipine. Thus, there's no enough safety data and efficacy data defined from the clinical study.

Also, many combination drugs of valsartaa and amlodipine are widely used in the market.

LGLS will compare the safety(adverse events especially the lower leg edema) and efficacy (blood pressure and pulse) of Levacalm and Valsartan/amlodipine combination drug from this study.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 19 with essential hypertension
* Those who meet the inclusion criteria, fall under any of the following 3 cases and determined by the investigator to be prescribed Levacalm or Valsartan/Amlodipine combination:

  1. those who can't maintain the blood pressure with the antihypertensive drug before.
  2. those who diagnosed to a hypertension stage 2.(DBP is higher than 160mmHg or SBP is higher than 100mmHg)
  3. those who fall under the following :cardiovascular disease, Cerebrovascular disease, chronic Renal disease, diabetes mellitus, peripheral vascular disease
* Those who were informed of the purpose, method, and effect etc. of this study and signed the informed consent form.

Exclusion Criteria:

1. Those who are included in the contraindication of study drug following the information for use of the product
2. Those who is/will be participated in other drug clinical trial
3. Those who adminitrated other antihypertensive drugs beside the levacalm or Valsartan/amlodipine combination drug.
4. Those who judged by the invesigator as ineligible for this clinical study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with essential hypertension
Sampling Method: Non-Probability Sample
Enrollment: 2001 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Safety of each group by observing the Adverse events especially detecting the incidence of lower leg edema and orthostatic hypertension by subject questionnaire. | 6month

SECONDARY OUTCOMES:
mean change of the blood pressure and pulse after administation of drug at 12week and 24week. | 12weeks, 24weeks
BP control rate | 12weeks, 24weeks
Responder rate | 12weeks, 24weeks
Evaluation of the changes in metabolic syndrome markers after treatment if the factors are available | 12weeks, 24weeks
Evaluation of cardiovascular risk | 12weeks, 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Keun Soo Bang, Study Director — LG Life Sciences
Locations (1):
- LG Life Science, Seoul, Jongno gu, South Korea